CLINICAL TRIAL: NCT00938106
Title: Implementation of Optimized Magnetic Resonance Image-guided Intra-uterine Brachytherapy in Cervical Cancer
Brief Title: Optimized Magnetic Resonance Brachytherapy (MR BT) in Cervix Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 08-0206-C
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Cervix Cancer
Keywords: Intra-uterine Brachytherapy; cervix cancer; Patients suitable for intra-uterine brachytherapy for invasive carcinoma of the cervix.
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- (MR BT) in Cervix Cancer (Experimental)
  Interventions: Radiation: optimised magnetic resonance image-guided intra-uterine brachytherapy

INTERVENTIONS:
Radiation: optimised magnetic resonance image-guided intra-uterine brachytherapy — Brachytherapy treatment will be planned based on the MRI test and will be individualized for each study participant,based on participant's cancer and body inside.Brachytherapy will be as an inpatient over 2-3 days. All other care will follow standard procedures.

SUMMARY:
Patients with cervix cancer usually require external radiation given to the whole pelvis then an internal radiation boost, also called brachytherapy, to treat any remaining tumour. Standard brachytherapy has been used successfully for many years, but does not take into account differences in the shape of the tumour or normal structures between patients. This study aims to implement individualized -optimized- brachytherapy, based on international recommendations. MR scanning with the intra-uterine applicator in place allows improved identification of residual tumour and normal structures, allowing brachytherapy to be individualized for each patient with the aim to reduce side-effects and improve outcome. Additionally, repeating MR scans during brachytherapy treatment will allow further assessment on motion of the applicator during treatment and the effect on radiation dose. Sexual health assessments aim to identify the relationship between sexual health and treatment effects.

DETAILED DESCRIPTION:
Pre-treatment: Prior to examination under anaesthesia and placement of the intra-uterine applicator, in addition to standard assessment of treatment toxicity, the patient may complete an optional Sexual Health assessment taking approximately 15 minutes. Following standard insertion of the intra-uterine applicator under general anaesthetic and planning MRI scan, there is an optional additional MRI scan taking an extra 30 minutes This extra scan will not affect the commencement of treatment planning as images from the planning scan will be transferred to the treatment planning system as soon as they are obtained. From the MRi planning scan, target and specific normal structures are contoured. An individual BT plan will be derived based on a standard plan to deliver dose within specified dose volume constraints.

During treatment: During inpatient BT optional MRI scans, each taking 15 minutes will be obtained in the period between treatment pulses once during each 24 hours of admission. The information from the additional MRI scans will not be used to alter or influence treatment.

Follow-up: Standard follow-up procedures will be followed, with the optional addition of the Sexual Health evaluation at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* ECOG performance status 0-2
* Histological confirmed carcinoma cervix
* Decision to treat with EBRT (+/- concurrent chemotherapy), and PDR BT
* Ability to comply with study protocol
* Patient informed consent

Exclusion Criteria:

* Unable to or unwilling to give informed consent
* Not suitable for intra-uterine brachytherapy
* Previous treatment for pelvic malignancy
* Previous pelvic radiotherapy
* Serious claustrophobia
* Previous history of metallic injury to the eye
* Non-removable implants contraindicated for MRI
* Cardiac pacemaker
* Other contraindication to MRI -Pregnancy, lactation or child-bearing potential without adequate contraception -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of clinical implementation of an effective and safe protocol for optimised MR image guided intra-uterine brachytherapy for cervix cancer. | 36 months

SECONDARY OUTCOMES:
Determine local control,overall survival,acute & late toxicity, & sexual health of patients treated with optimised intra-uterine BT. Evaluate stability of the intra-uterine applicator during BT. Evaluate dose homogeneity of BT for cervix cancer. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Milosevic, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Toronto, Ontario, Canada